CLINICAL TRIAL: NCT01196780
Title: MabThera Post Marketing Observational Study in TNF-IR Patients to Assess Efficacy and Safety of REPeated Courses in routinE ClinicAl pracTice
Brief Title: An Observational Study of MabThera/Rituxan (Rituximab) in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Anti-TNF Therapy (REPEAT)
Status: Terminated | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25228
Record Dates: First submitted 2010-09-06; First posted 2010-09-08 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will assess the efficacy and safety of MabThera/Rituxan (Rituximab) in patients with active rheumatoid arthritis who have had an inadequate response or are intolerant to anti-TNF therapy. Data will be collected from patients initiated on MabThera/Rituxan therapy according to standard of care in routine clinical practice. For each patient data will be collected for 92 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active Rheumatoid Arthritis
* Inadequate response to anti-TNF
* Eligible for MabThera/Rituxan therapy according to physician's decision

Exclusion Criteria:

* According to Summary of Product Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an inadequate response to prior anti-TNF therapy
Sampling Method: Probability Sample
Enrollment: 1240 (Actual)
Dates: Start 2010-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Efficacy: Change in Disease Activity Score - erythrocyte sedimentation rate (DAS28 - ESR) | from baseline to Week 92

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bucharest, Romania